CLINICAL TRIAL: NCT01514058
Title: A Prospective, Randomized Study Evaluating the Effect of Biliary Stenting on EAU-FNA in Patients With Suspected Malignant Biliary Obstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: new clinical strategies have rendered the question posed by this study less relevant
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00018166; CCCWFU 01711 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-01-12; First posted 2012-01-20 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Jaundice
MeSH Terms: conditions — Jaundice | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-FNA First (Active Comparator): Patients will undergo EUS-FNA first, followed by ERCP with biliary stenting (using a plastic stent).
  Interventions: Procedure: EUS-FNA first, followed by CRCP with bilinary stenting
- ERCP with stent placement first (Active Comparator): Patients will undergo ERCP with stent placement first, followed by EUS-FNA.
  Interventions: Procedure: ERCP with stent placement, followed by EUS-FNA

INTERVENTIONS:
Procedure: EUS-FNA first, followed by CRCP with bilinary stenting — EUS-FNA first, followed by CRCP with bilinary stenting (using a plastic stent)
  Arms: EUS-FNA First
Procedure: ERCP with stent placement, followed by EUS-FNA — ERCP with stent placement, followed by EUS-FNA
  Arms: ERCP with stent placement first

SUMMARY:
Patients who present with obstructive jaundice due to a malignant stricture often undergo a battery of tests for diagnosis, treatment options, and prognosis. An endoscopic retrograde cholangiopancreatography (ERCP) is often performed with biliary stent placement for symptom relief as well as brushings for cytology. An endoscopic ultrasound is performed as well for fine needle aspiration (FNA) of the pancreas to aid in diagnosis. However, since EUS is not available at many centers, patients often undergo an initial ERCP procedure with stent placement (which is more widely available) prior to referral for EUS. It has been reported that biliary stents can disturb EUS visualization due to inflammation, acoustic shadowing, and pneumobilia which may lessen the accuracy of diagnosis.1 The cytological yield from the EUS with FNA procedure may also be compromised in patients with biliary stents. As such, diagnosis and treatment options may be delayed. One retrospective study of 65 subjects showed a significant difference in the number of correctly staged pancreatic head cancers (mainly T stage) in patients without stents versus those with biliary stents (85% vs 47%).2 A second retrospective study concluded that tissue diagnosis is not influenced in patients with stents placed greater than 24 hours before the EUS; however, patients with stents placed just prior to the EUS (less than 24 hours) were more likely to have indeterminate results.1 Although the findings are suggestive, the studies are limited by their retrospective design and these questions have not yet been addressed in a prospective study.

Both procedures require anesthesia, and when performed sequentially in the same setting, the duration of anesthesia is prolonged. This is concerning for the patient since complications may theoretically increase with prolonged anesthesia. However, a retrospective review at a tertiary referral center showed that combined EUS and ERCP yielded a complication rate no higher than that of the component procedures.3

At our institution, the current practice is to sequentially perform both EUS and ERCP in the same setting for patients with suspected malignant biliary obstruction. Typically, EUS-FNA is performed first, followed by ERCP.

Hypothesis We hypothesize that performing ERCP with biliary stenting immediately prior to EUS-FNA will decrease the diagnostic yield of EUS-FNA and diminish the ability of EUS to accurately stage pancreas tumors. Conversely, performing EUS-FNA prior to ERCP will increase biliary cannulation time and increase success rate.

The objectives of this study are as follows:

1. Determine the diagnostic yield of EUS-FNA (for diagnosis of cancer vs benign process) when performed either immediately before or after ERCP with biliary stenting (primary outcome)
2. Determine the ability of EUS to accurately stage pancreatic masses (T and N staging) when performed either immediately before or after ERCP with biliary stenting (secondary outcome) in comparison to the gold standard of surgical pathology post resection or in comparison to CT findings (in those patients who are not surgical candidates)
3. Determine the biliary cannulation time (the time it takes to successfully pass a wire into the common bile duct from the start of the procedure) and success rate of placing a biliary stent during ERCP when performed either immediately before or after EUS-FNA (secondary outcome)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to review and sign informed consent.
* Subjects must require biliary stenting for the relief of their symptoms as well as FNA biopsy for proper diagnosis.
* Suspected mass should be located in the head, uncinate, or neck of the pancreas.

Exclusion Criteria:

* Cannot give and sign informed consent.
* The suspected mass is located in the body or tail of the pancreas.
* The patient may be a candidate for palliative biliary stenting (in which a metal stent would be placed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Cytological yield (adequate versus inadequate for diagnosis) of EUS-FNA prior to stent placement vs post stent placement | 1 day
  Cytological yield will be defined by the ability of the pathologist to render a diagnosis based on the material supplied to them during the procedure (adequate vs inadequate tissue to make a diagnosis of malignant vs benign disease).

CONTACTS AND LOCATIONS:
Overall Officials: John A Evans, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States